CLINICAL TRIAL: NCT00729131
Title: Functional Implications of TNF
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Michael Foster, Professor, National Institute of Environmental Health Sciences (NIEHS)
Other Study IDs: 00008547
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Bronchitis
Keywords: Ozone, TNF, TNF promoter polymorphism, airway hyperresponsiveness.
MeSH Terms: conditions — Bronchitis; Respiratory Hypersensitivity | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage specimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Control group: subjects are homozygotic for major allele for TNF-308 promoter polymorphism.
  Interventions: Drug: Etanercept inhibition of ozone-induced airway hyper-responsiveness.
- B: Case Group: subjects are homozygotic or heterozygotic for minor allele of TNF-308 promoter polymorphism.

INTERVENTIONS:
Drug: Etanercept inhibition of ozone-induced airway hyper-responsiveness. — Single dosage of etanercept(50 mg, subcutaneous) given 2 days prior to a laboratory ozone exposure.
  Other Names: Only a single group of subjects, known to demonstrate airway hyperresponsiveness at 20 hr post exposure to ozone will be studied in the; intervention.
  Groups: A

SUMMARY:
The research plan proposes to develop translational studies in humans that will identify host susceptibility factors that confer vulnerability to the prototypal air pollutant, ozone. Ozone is a ubiquitous urban air pollutant and associated with increased emergency room visits, and co-associates with other air pollutants, to increase mortality in high risk groups (cardio-pulmonary disease) of the population.The results will have significant impact upon and aid in understanding mechanisms of pro-oxidant lung injury, airway hyperresponsiveness, and adverse health effects, that occur during and following exposure to inhalable airborne irritants.

DETAILED DESCRIPTION:
Exposure of the airways to air toxins initiates transient and reversible airway injury to both adults and young children. Repetitive exposures of children residing within high oxidant communities leads to impairment of lung growth and pulmonary function, and remodeling of airway epithelial tissues is also suggested to occur. In the completely normal/healthy airway, exposure to ozone (O3), a ubiquitous urban air pollutant, induces an inflammatory response that is characterized by increases in epithelial permeability, neutrophilic infiltration, and bronchial hyperreactivity. Inhalation by humans of the pleiotropic pro-inflammatory cytokine tumor necrosis factor (Tnf) leads to the development of nearly identical responses: hyperresponsiveness of the bronchial airway (AHR), and neutrophil influx. Using controlled exposure to O3 in a laboratory setting, we have recently established a link between a genetic single nucleotide polymorphism (SNP) of TNF gene (-308) and the development of AHR to methacholine within a 24 h time frame, post exposure to O3. In a healthy human study group (n=137) the presence of a common TNF (-308) SNP was found to confer susceptibility to an ambient concentration of O3 (220 ppb, and frequently attained in many cities of the US during the summer months): stratified for ethnicity, Caucasian subjects who were homozygotic (A/A) or heterozygotic (G/A) for the minor allele of the TNF (-308) SNP were 2-times as likely to develop sensitivity to methacholine after O3 as compared to subjects with the wild-type, major allele (G/G) haplotype.

Literature reports suggest that the TNF(-308) polymorphism associates with increased TNF gene transcription and increased Tnf cytokine production. However, the functional significance of this common TNF polymorphism remains uncertain; and moreover, the functional implications of the TNF(-308) polymorphism in the lung remain undeveloped. We hypothesize that subjects either homozygotic (A/A) or heterozygotic (G/A) for the minor allele of the TNF(-308) promoter polymorphism, will demonstrate enhancement in phenotypic responses to O3 including: increased cellular inflammation and secretion of pre-inflammation cytokines, enhanced activation of resident alveolar macrophages, and altered bronchial sensitivity, leading to AHR.

Our research plan is designed to mechanistically investigate the interaction between host factors of humans and exposure to the prototypal air pollutant, ozone. The research plan will expand upon, and enable, a clear assignment of the functional contribution of a common SNP of TNF gene to the initiation of airway hyperresponsiveness, a cardinal feature of inflammatory airway disease.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* subjects with current or past smoking history, acute respiratory illness within six weeks of the study, and significant non-pulmonary disease as determined by the investigator, pregnancy, age <18 or >35 yr, or inability to understand the protocol. Subjects will be requested to refrain from anti-histamines, nonsteroidal anti-inflammatory agents, and supplemental vitamins, e.g. C and E, for 1 week prior to, and during lab visits for exposures and follow-up measures.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy non-smokers (18-35 yr) will be recruited from the Duke campus and local community; 50% will be women. Subjects will have a clinical history and lung function screening at protocol entry. Female subjects of childbearing age will have pregnancy testing. We will only recruit subjects with a normal body habitus as an increased BMI may modify sensitivity to O3. Subjects will have lung volumes within predicted normal, and FEV1, and FEF25-75, within range of predicted, and methacholine response less than the mean Mch PC20 dose for non-asthmatic population in our human inhalation laboratory. Atopic status of study subjects will be determined by lack of positive skin test by prick technique (using panel of antigens common to central NC) and without seasonal or perennial allergic symptoms.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
biologic response to ozone exposure: bronchoalveolar lavage fluid analyzed for inflammatory cytokines, cell differentials, and activated alveolar macrophages. | Lung lavage evaluated 20 hr post-exposure to ozone.

SECONDARY OUTCOMES:
Alveolar macrophages (collected in lung lavage fluid) will be studied ex vivo for activation state and pro-inflammatory cytokine secretion. | 20 hr post-exposure to ozone.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States